CLINICAL TRIAL: NCT00347126
Title: Efficacy and Safety of a Systematic Switch From Latanoprost to Travoprost in Patients With Glaucoma
Brief Title: Results of Mass Switch From Latanoprost to Travoprost
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Other Study IDs: R463/12/2006
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Glaucoma
Keywords: Glaucoma; Latanoprost; Travoprost; Intraocular pressure; Hyperemia
MeSH Terms: conditions — Glaucoma; Hyperemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Prostaglandin analogs are a leading class of glaucoma drugs with a proven safety and efficacy for controlling IOP. They include latanoprost, bimatoprost, travoprost and unoprostone. Recently, the Singapore National Eye Center (SNEC) awarded a tender for prostaglandin analogues to Alcon, the manufacturer of travoprost. Since then, all subsidized patients previously treated with latanoprost were systematically switched to travoprost and this process will continue for the rest of this year. In this study, we propose to prospectively study the efficacy and safety of switching from latanoprost to travoprost in a large series of glaucoma patients at SNEC. A total of 372 consecutive patients being switched from latanoprost to travoprost will be followed up for 12 weeks following the switch. In addition to intraocular pressure, the safety and tolerability (with particular emphasis on hyperemia) of travoprost will be examined.

DETAILED DESCRIPTION:
Aims:

1. To assess the feasibility of switching a large group of patients on treatment with latanoprost to travoprost.
2. To assess the efficacy and safety of travoprost compared to latanoprost after the switch.

Intraocular pressure (IOP) is currently the only proven modifiable risk factor in the management of glaucoma.1 Either medical or surgical management can achieve the control of IOP. Prostaglandin analogs are the newer class of drugs among the various topical ocular hypotensive medications, with a proven safety and efficacy for controlling IOP.2 Their potency and once a day dosing and lower incidence of systemic side effects have made them popular for use as monotherapeutic and first-line agents. They include latanoprost, bimatoprost, travoprost and unoprostone. All of them have a similar molecular structure and they work by increasing the aqueous drainage via trabecular meshwork and the uveoscleral pathway.3 It has been shown that the efficacy of latanoprost, bimatoprost and travoprost in reducing IOP in ocular hypertension and primary open angle glaucoma is comparable.4 Conjunctival hyperemia is one of the most common ocular side effects. There has been a reported higher incidence of hyperemia with bimatoprost and travoprost as compared to latanoprost.4 However, this hyperemia is usually benign and usually abates as the drug is used long term. The incidence of discontinuation of therapy due to hyperemia is very low and not different among the various prostaglandins.5 Among the prostaglandin analogues, latanoprost has been the market leader in Singapore for the past few years. However, the Singapore National Eye Center (SNEC) pharmacy recently accepted tenders from various drug companies for prostaglandin analogs. Alcon, the manufacturer of travoprost was awarded the tender. Since then, all subsidized patients previously treated with latanoprost were systematically switched to travoprost and this process will continue for the rest of this year. The switch is a systematic switch and is not based on intolerance or poor response to latanoprost.

To date, there has been a single report regarding the feasibility and efficacy of a mass switch from latanoprost to bimatoprost.5 The study reported a high switch rate and good IOP control with minimal switch back. However, similar data on switching from latanoprost to travoprost is lacking. In this study, we propose to prospectively study the efficacy and safety of switching from latanoprost to travoprost in a large series of glaucoma patients at SNEC. A total of 372 consecutive patients being switched from latanoprost to travoprost will be followed up for 12 weeks following the switch. In addition to IOP, safety and tolerability (with particular emphasis on hyperemia) of travoprost will be examined.

References:

1. Leske MC, Heijl A, Hussein M et al. Factors for glaucoma progression and the effect of treatment: the early manifest glaucoma trial. Arch Ophthalmol. 2003 Jan;121(1):48-56.
2. Alexander CL, Miller SJ, Abel SR. Prostaglandin analog treatment of glaucoma and ocular hypertension. Ann Pharmacother. 2002 Mar;36(3):504-11.3.
3. Eisenberg DL, Toris CB, Camras CB. Bimatoprost and travoprost: a review of recent studies of two new glaucoma drugs. Surv Ophthalmol. 2002 Aug;47 Suppl 1:S105-15.
4. Parrish RK, Palmberg P, Sheu WP; XLT Study Group. A comparison of latanoprost, bimatoprost, and travoprost in patients with elevated intraocular pressure: a 12-week, randomized, masked-evaluator multicenter study. Am J Ophthalmol. 2003 May;135(5):688-703.
5. Law SK, Song BJ, Fang E, Caprioli J. Feasibility and efficacy of a mass switch from latanoprost to bimatoprost in glaucoma patients in a prepaid Health Maintenance Organization. Ophthalmology. 2005 Dec;112(12):2123-30.

ELIGIBILITY:
Inclusion Criteria:

1. Patients on treatment with latanoprost for at least 12 weeks; patients who are on additional beta-blockers topically will also be eligible.
2. Written informed consent. -

Exclusion Criteria:

1. Patients on 3 or more topical medications.
2. Recorded history of intolerance to travoprost.
3. Recorded history of inefficacy of travoprost in controlling IOP.
4. Patients on any additional topical medication other than beta-blockers.
5. History of non-compliance.
6. Involvement in any other concomitant study. -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients on treatment with latanoprost who are switched to travoprost therapy
Sampling Method: Non-Probability Sample
Enrollment: 372 (Estimated)
Dates: Start 2006-04; Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tin Aung, FRCS, PhD, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore